CLINICAL TRIAL: NCT07373756
Title: Effectiveness Of Aspirin In The Prevention Of Preeclampsia In High Gestosis Scored Women Attending Tertiary Level Hospital In Kathmandu: A Randomized Controlled Trial
Brief Title: Randomized Controlled Study to Compare Efficacy of Aspirin 75mg and 150mg In the Prevention of Preeclampsia In High Risk Pregnant Women
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Sunita Pun (Other)
Responsible Party: Sponsor-Investigator, Dr. Sunita Pun, Pricipal Investigator, Tribhuvan University, Nepal
Organization: Tribhuvan University, Nepal (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 599/2025
Record Dates: First submitted 2026-01-14; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy Induced Hypertension (PIH)
Keywords: hypertension, preeclampsia, aspirin
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension; Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 75mg Aspirin Arm (Experimental): Interventional
  Interventions: Drug: Aspirin
- 150mg Aspirin Arm (Active Comparator): Interventional
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — This interventional study is being doe in pregnant women after calculationg their Gestosis score and if Gestosis score of 3 or more, they will be randomised into aspirin 75mg and aspirin 150mg in the ratio 1:1. After their delivery, the result will be recorded as to whether preeclampsia had been prevented.

SUMMARY:
Preeclampsia in pregnancy is a dreaded complication which has both fetal and maternal adverse outcomes. Studies and WHO have advocated that this complication can be prevented by Aspirin. However which dose is more effective in preventing preeclampsia, whether 75mg or 150mg, will be known from this study.

DETAILED DESCRIPTION:
Preeclampsia is a leading cause of maternal and perinatal morbidity and mortality worldwide, particularly in low- and middle-income countries. It is a multisystem disorder of pregnancy characterized by new-onset hypertension after 20 weeks of gestation, often accompanied by proteinuria or evidence of end-organ dysfunction. The pathophysiology of preeclampsia involves abnormal placentation, endothelial dysfunction, increased platelet activation, and an imbalance between vasoconstrictive and vasodilatory prostaglandins.

Low-dose Aspirin (acetylsalicylic acid) has been shown to reduce the risk of preeclampsia through irreversible inhibition of cyclooxygenase-1 (COX-1), resulting in reduced thromboxane A2 production, decreased platelet aggregation, and improved uteroplacental perfusion. International guidelines recommend prophylactic low-dose Aspirin for pregnant women at high risk of preeclampsia; however, there is ongoing debate regarding the optimal dose. Both 75 mg and 150 mg doses are currently used in clinical practice, but comparative evidence in South Asian populations, including Nepal, remains limited.

This investigator-initiated, non-commercial randomized controlled trial is designed to compare the effectiveness and safety of Aspirin 75 mg versus Aspirin 150 mg once daily for the prevention of preeclampsia in pregnant women identified as high risk based on a high gestosis score. The study is conducted at a tertiary-level teaching hospital in Kathmandu, Nepal.

Participants will be enrolled during early pregnancy and randomized in a 1:1 allocation ratio to receive either Aspirin 75 mg or Aspirin 150 mg orally once daily. Randomization will be generated using a computer-based random sequence with block randomization to ensure balance between treatment groups. Allocation concealment will be achieved using sequentially numbered, opaque, sealed envelopes prepared by an independent individual not involved in participant recruitment or outcome assessment.

Due to the difference in tablet strength, the trial is open-label. To minimize bias, all participants will receive identical standard antenatal care according to institutional and national guidelines, and outcome assessment will follow predefined diagnostic criteria. Data analysis will be conducted by investigators blinded to treatment allocation.

The investigational product will be administered from enrollment until 36 weeks of gestation or delivery, whichever occurs earlier. Participants will be advised to take the study medication once daily, preferably at bedtime. The intervention will not replace or interfere with routine antenatal care, and all co-interventions will be documented.

Participants will be followed throughout pregnancy during scheduled antenatal visits. Follow-up assessments will include monitoring of blood pressure, urine protein testing, evaluation for clinical features of hypertensive disorders of pregnancy, and assessment of adherence to the study medication. Compliance will be evaluated using participant self-reporting and pill counts.

Safety monitoring is an integral component of the study. Adverse events and serious adverse events will be actively monitored throughout the study period. A predefined safety monitoring and Serious Adverse Event (SAE) management plan is in place, consistent with ICH Good Clinical Practice (GCP) guidelines and the Ethical Guidelines for Health Research in Nepal. Any SAE will be promptly managed according to standard institutional clinical protocols, with immediate discontinuation of the investigational product if indicated. Causality assessment will be performed using the WHO-UMC criteria, and SAEs will be reported to the Institutional Review Committee and the Nepal Health Research Council Ethical Review Board within required timelines.

An independent Data Safety Monitoring Board (DSMB) will periodically review accumulated safety data and provide recommendations regarding study continuation, modification, or termination based on safety considerations.

Study data will be collected using structured case report forms and entered into a secure electronic database. Participant confidentiality will be maintained by assigning unique study identification numbers. Identifiable information will be stored separately from clinical data and accessed only by authorized study personnel. Data quality assurance measures include regular data checks, monitoring, and adherence to standard operating procedures.

The study aims to generate locally relevant evidence regarding the optimal prophylactic dose of Aspirin for the prevention of preeclampsia in high-risk pregnant women in Nepal. Given the low cost, wide availability, and established safety profile of low-dose Aspirin, the findings may inform clinical practice and contribute to improved maternal health outcomes in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* • All pregnant women with Gestosis score of 3 or more who consents for the study and aged 18 years and above.

Exclusion Criteria:

* • Known hypersensitivity to aspirin, uncontrolled asthma with NSAID sensitivity

  * Bleeding disorders, platelet dysfunction, thrombocytopenia, anticoagulant use, active peptic ulcer, history of GI bleed, severe hepatic/ renal disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 86 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Preeclampsia | 1 year (After the time of randomization till delivery)
  Preeclampsia will be assessed during routine antenatal visits and at delivery by trained obstetric clinicians. Blood pressure will be measured using a calibrated sphygmomanometer with the participant in a seated position after adequate rest. Hypertension will be defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg recorded on two occasions at least 4 hours apart after 20 weeks of gestation. Proteinuria will be assessed using urine dipstick testing (≥1+) or 24-hour urine protein estimation (≥300 mg). In the absence of proteinuria, preeclampsia will be diagnosed based on hypertension with evidence of maternal end-organ dysfunction. The incidence of preeclampsia will be recorded after the the time of randomization until delivery .